CLINICAL TRIAL: NCT04949971
Title: Peking University Third Hospital
Brief Title: A Comparative Study of High and Low Tidal Volume in Preventing Hypoxemia in Patients With Mechanical Ventilation After Cervical Spinal Cord Injury
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: LM2020353
Record Dates: First submitted 2021-06-29; First posted 2021-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2020-08

CONDITIONS: Cervical Spinal Cord Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High volume group: The tidal volume of the exposed group was 10ml/kg ideal body weight.
- Low volume group: The tidal volume of the non-exposed group was 6ml/kg ideal body weight
  Interventions: Behavioral: High volume group

INTERVENTIONS:
Behavioral: High volume group — Thea High tidal volume of the exposed group was 10ml/kg ideal body weight
  Other Names: Low volume group
  Groups: Low volume group

SUMMARY:
This study in order to best tidal volume mechanical ventilation in patients with cervical spinal cord injury (sci) as the research point, through higher low volume Settings to find the difference of two groups of patients to prevent the incidence of hypoxemia, to find suitable Settings, tidal volume in patients with lower mechanical ventilation in patients with cervical spinal cord injury (sci) the incidence of pulmonary complications, live less intensive care unit (ICU).

ELIGIBILITY:
Inclusion Criteria:

* All critically ill adult patients with cervical spinal cord injury who require mechanical ventilation and informed consent to be admitted to the Department of Critical Care Medicine of Peking University Third Hospital were selected by the subjects or their close relatives to enter the clinical study.

Exclusion Criteria:

* previous chronic obstructive pulmonary disease, diagnosis of acute respiratory distress syndrome at admission, presence of pneumothorax at admission, subjects or close relatives who refused to participate in the study, and non-signed informed consent."

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ① Above the age of 18;
  ② Patients with cervical spinal cord injury requiring mechanical ventilation admitted to hospital.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of hypoxemia | during machinical ventilation
  The oxygenation index is less than 300

CONTACTS AND LOCATIONS:
Locations (1):
- Xuelei, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided